CLINICAL TRIAL: NCT06731673
Title: Heat Shock Protein 47: A Novel Biomarker of Thrombosis Risk
Brief Title: Heat Shock Protein 47 in Thrombosis
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Max Planck Institute of Biochemistry (Unknown); Deutsches Herzzentrum der Charité, Berlin (Unknown)
Responsible Party: Sponsor
Other Study IDs: HSP47
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2024-12

CONDITIONS: Venous Thromboembolism (VTE); Acute Myocardial Infarction With ST Segment Elevation; Stroke (in Patients With Atrial Fibrillation)
Keywords: HSP47; Heat Shock Protein 47; Biomarker; Novel biomarker; Trombosis; VTE; AMI; Stroke
MeSH Terms: conditions — Venous Thromboembolism; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Venous thromboembolism: Patients with acute deep vein thrombosis diagnosed on UL or pulmonary embolism diagnosed on CTA. >18 years of age. 120 patients in total.
- Acute myocardial infarction: With ST segment elevation on ECG and confirmed culprit lesion on coronary angiography. >18 years of age. 50 patients in total.
- Stroke: Stroke confirmed on MRI and diagnosis of atrial fibrillation. >18 years of age. 50 patients in total.
- Healthy participants: No known or prior diseases, no medication. >18 years of age. 120 in total.

SUMMARY:
The goal of this observational study is to learn if the novel biomarker Heat shock protein 47 (HSP47) can be used as a prognostic marker for vascular disease in people with acute venous thromboembolism (VTE), myocardial infarction (AMI) or ischaemic stroke compared to healthy volunteers. The main questions it aims to answer are:

1. Are platelet levels of HSP47 higher in patients with acute VTE, AMI or stroke, compared to healthy volunteers.
2. Does platelet levels of HSP47 remain elevated in patients with acute thrombotic events compared to healthy volunteers at 3 and 12-months of follow-up.
3. Are platelet levels of HSP47 postively associated with platelet function and negatively associated with fibrinolytic capacity in patients with an acute thrombotic event.

Participants with VTE, AMI or stroke will be giving a blood sample at diagnosis and again after 3 and 12 months of follow-up. Healthy volunteers will be giving a blood sample once.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Informed consent

VTE group:

* Deep vein thrombosis confirmed on ultrasonography OR
* Pulmonary embolism confirmed on computed tomography angiography (CTA)

AMI group:

* ST-segment elevation on electrocardiogram (ECG) AND
* Culprit lesion(s) on coronary angiography

Stroke group:

* Stroke confirmed on magnetic resonance imaging AND
* Atrial fibrillation (Detected on ECG, telemtry or Holter monitoring) AND
* Stroke localisation classic for AFib: cortical, cerebellar, brainstem or subcortical >1.5 cm in diameter

Healthy group:

- Healthy

Exclusion Criteria:

* <18 years of age
* no informed consent
* Known haematological disorders
* Active haematological malignancy
* Severe renal insufficiency defined as eGFR <15 or dialysis

VTE - Pulmonary embolism incidentally detected by CTA conducted for purposes unrelated to pulmonary embolism assessment without concomitant DVT

AMI

* Coronary dissection
* Takotsubo cardiomyopathy

Stroke

- Stroke from other causes, e.g. findings pointing towards large vessel disease

Healthy

* Known acute or chronic disease
* Prior VTE, AMI, stroke or other thromboembolic event

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited at Aarhus University Hospital at the department of Cardiology (AMI, VTE), Neurology (Stroke) and Radiology (VTE) and at the Blood Bank (Healthy volunteers).
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Platelet levels of heat shock protein 47 (HSP47) in patients with thrombosis compared to healthy controls | From enrollment to end of follow-up at 12 months after enrollment. At 3 time points.
  The level of HSP47 on platelets will be measured in a bloodsample. It will be measured using proteomics and flow cytometry.

SECONDARY OUTCOMES:
Changes in platelet levels of HSP47 over time in patients with thrombosis | From enrollment to 12 months of follow-up. Measured at 3 time points.
  The level of HSP47 on platelets will be measured in a bloodsample. It will be measured using proteomics and flow cytometry.
Platelet levels of HSP47 in association to platelet function | From enrollment to 12 months of follow-up. Measured at 3 time points.
  The level of HSP47 on platelets will be measured in a bloodsample. It will be measured using proteomics and flow cytometry. Platelet function will be assessed by platelet aggregation and activation using impedance aggregometry and flow cytometry.
Platelet levels of HSP47 in association to fibrinolytic capacity | From enrollment to 12 months of follow-up. Measured at 3 time points.
  The level of HSP47 on platelets will be measured in a bloodsample. It will be measured using proteomics and flow cytometry. Fibrinolytic capacity will be assessed by ROTEM (R) tPA methods established in our lab, and by plasma fibrinolysis analyses.

CONTACTS AND LOCATIONS:
Locations (2):
- Aarhus University Hospital, Aarhus, Central Region, Denmark
- Deutsches Herzzentrum de Charité, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thienel M, Muller-Reif JB, Zhang Z, Ehreiser V, Huth J, Shchurovska K, Kilani B, Schweizer L, Geyer PE, Zwiebel M, Novotny J, Lusebrink E, Little G, Orban M, Nicolai L, El Nemr S, Titova A, Spannagl M, Kindberg J, Evans AL, Mach O, Vogel M, Tiedt S, Ormanns S, Kessler B, Dueck A, Friebe A, Jorgensen PG, Majzoub-Altweck M, Blutke A, Polzin A, Stark K, Kaab S, Maier D, Gibbins JM, Limper U, Frobert O, Mann M, Massberg S, Petzold T. Immobility-associated thromboprotection is conserved across mammalian species from bear to human. Science. 2023 Apr 14;380(6641):178-187. doi: 10.1126/science.abo5044. Epub 2023 Apr 13. PMID 37053338